CLINICAL TRIAL: NCT02645474
Title: Is PECS Block Equivalent to Paravertebral Block in Preventing Postoperative Pain After Breast Surgery? A Randomized, Controlled, Double-blind, Multicenter Trial
Brief Title: Is PECS Block Equivalent to Paravertebral Block in Preventing Postoperative Pain After Breast Surgery?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ospedale Regionale Bellinzona e Valli (Other)
Responsible Party: Principal Investigator, Andrea Saporito, Andrea Saporito MD, Ospedale Regionale Bellinzona e Valli
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PECS
Record Dates: First submitted 2015-12-29; First posted 2016-01-01 (Estimated); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Other Acute Postoperative Pain
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paravertebral block with ropivacaine (Active Comparator): Patients are treated with an older technique (paravertebral block with ropivacaine), somehow established in treating pain after breast surgery. This technique has been shown to be effective but has an intrinsic risk of iatrogenic pneumothorax and is considered technically demanding.
  Interventions: Procedure: Paravertebral block with ropivacaine; Drug: Ropivacaine
- PECS block with ropivacaine (Experimental): Patients are treated with PECS block, which has been already adopted in common clinical practice as an alternative to paravertebral block for postoperative pain treatment after breast surgery. This technique is thought to be somehow simpler to perform and safer with regard to pneumothorax, however no studies have been done yet to statistically compare the two blocks with regard to safety and effectiveness.
  Interventions: Procedure: PECS block with ropivacaine; Drug: Ropivacaine

INTERVENTIONS:
Procedure: PECS block with ropivacaine — Local anesthetic (ropivacaine 0.5%, total volume 30 ml) is infiltrated in between the fasciae of serratus and minor pectoralis muscles under ultrasound guidance.
  Other Names: Pectoral muscles sheath block
  Arms: PECS block with ropivacaine
Procedure: Paravertebral block with ropivacaine — Local anesthetic (ropivacaine 0.5%, total volume 20 ml) is infiltrated in the paravertebral block at T4 level under ultrasound guidance.
  Other Names: PVB
  Arms: Paravertebral block with ropivacaine
Drug: Ropivacaine — Amidic local anesthetic standardly used for nerve block and infiltration
  Other Names: Naropine

SUMMARY:
Two regional anesthesia techniques already in use in common clinical practice -paravertebral block and pectoral nerve block (PECS block) are compared in a randomized, double-blind, multicenter, controlled, non-inferiority trial, in order to compare their success rate in patients udergoing breast surgery.

DETAILED DESCRIPTION:
Aim of the study is to compare paravertebral block and PECS block success rate in patients undergoing elective breast surgery (mastectomy or quadrantectomy) with a combined anesthesia technique.

Primary outcome is block success rate defined as a VAS score of 30 or less in PACU and at 6, 12 and 24 hours after surgery. Secondary outcomes are: rescue opioids requirement; incidence of procedure related complications; incidence of postoperative side-effects; patients' quality of life level during the first 24 postoperative hours; patients' satisfaction.

A prospective, randomized, controlled, double-blinded, non-inferiority trial was designed in order to compare paravertebral block and PECS block with regard to block success over the first 24 hours postoperatively in patients undergoing mastectomy or quadrantectomy procedures with a combined anesthesia technique.

Inclusion criteria: adult patients, ASA class 1 to 3, scheduled for elective mastectomy or quadrantectomy. Exclusion criteria: patients refusal, contraindication to regional anaesthesia (coagulopathies, concurrent anticoagulant therapy, allergy to local anaesthetics, infection at puncture site).

After written informed consent, patients will be randomized into two cohorts, the first being treated with a paravertebral block, while the second with a PECS block. Both procedures will be standardized with regard to injection technique, local anaesthetic drug and volume and performed under ultrasound real-time guidance. Both groups will undergo the regional anesthesia technique after induction of general anaesthesia to be blinded with regard to the type of block. This will be standardized as well, according to our centers current clinical practice. Postoperative pain will be than measured on a validated visual analogue scale (VAS 0-100) in the recovery room and periodically after discharge to the ward until 24 hours postoperatively. Rescue opioids requirement will be recorded. Eventual procedural complications occurred will be recorded as well as postoperative side effects. A questionnaire about patients' satisfaction and quality of life during the first 24 postoperative hours will be filled in for every patient. Data collected will be initially inserted in a form and subsequently collected, pooled and anonymously registered in an electronic data base.

A sample size calculation has been preliminary performed with regard to the primary outcome. A 20% difference in the blocks success rate (defined as a postoperative pain on VAS scale of 30 or less) will be considered as clinically significant.

In our practice, paravertebral block is the current gold standard and it is associated on average to a 50% mean value on VAS scale during the first 48 postoperative hours. PECS block will be thus compared to this standard of care. A total of 39 patients per arm will be required (95% confidence interval). Accounting for a 10% drop-out rate, we will include 43 patients per arm.

Pain levels will be measured as medians and interquartile ranges. Statistical analysis will be performed using Student t-test for normally distributed variables while Mann-Whitney test was applied to non-normally distributed variables.

This study will be conducted in compliance with the protocol, the current version of the Declaration of Helsinki, the ICH-GCP or ISO EN 14155 (as far as applicable) as well as all national legal and regulatory requirements.

ELIGIBILITY:
Inclusion Criteria:

* adult patients
* ASA class 1 to 3 patients
* patients scheduled for elective breast mastectomy or quadrantectomy

Exclusion Criteria:

* patients' refusal
* contraindication to regional anaesthesia (coagulopathies, concurrent anticoagulant therapy, allergy to local anaesthetics, infection at puncture site)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Success rate (measured via visual analogue scale) | 24 hours after surgery
  Changes in postoperative pain level of intensity over time will be measured via visual analogue scale (on a 0 to 100 scale, where 0 means no pain and 100 stands for the maximum pain ever experienced). Patients in both groups will be asked to rate their postoperative pain levels at fixed intervals, i.e. in the postoperative anesthesia care unit and once in the ward at 6, 12, 24 hours after surgery

SECONDARY OUTCOMES:
Safety (incidence of complications) | 24 hours after surgery
  Safety will be assessed as incidence of complications in the two groups over the first 24hours. Complications monitored will be: clinical signs of pneumothorax, inadvertent vascular puncture, local anesthetic toxicity
Patients' satisfaction (subjective perception of the experience on a 0 to 100 scale) | 24 hours after surgery
  Patients will be asked to rate their satisfaction with regard to procedural pain and subjective perception of the experience on a 0 to 100 scale

CONTACTS AND LOCATIONS:
Overall Officials: Luciano Anselmi, MD, Study Chair — Ospedale Regionale di Bellinzona e Valli
Locations (1):
- Ospedale Regionale di Bellinzona e Valli, Bellinzona, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dossi R, Tasciotti E, van Sander K, Maino P, Reyes Lozano V, Saporito A, Koetsier E. Comparison of Pectoral Nerve and Paravertebral Blocks for Postoperative Pain Management in Breast Surgery: A Multicentre Randomised Double-Blind Trial. J Breast Cancer. 2025 Aug;28(4):268-279. doi: 10.4048/jbc.2025.0060. PMID 40887728